CLINICAL TRIAL: NCT03446625
Title: Resveratrol as a Preventive Treatment of Ovarian Hyperstimulation Syndrome
Brief Title: Resveratrol as a Preventive Treatment of OHSS
Acronym: RES-OHSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, MD, IVI Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1401-MAD-004-IO
Record Dates: First submitted 2017-01-12; First posted 2018-02-27 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2018-08

CONDITIONS: Infertility
Keywords: resveratrol; OHSS; PCOS
MeSH Terms: conditions — Infertility | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resveratrol (Experimental): Resveratrol will be administered orally at the dose of 2 g/day for 9 days, starting on the day of ovulation triggering.
  Interventions: Drug: Resveratrol; Drug: Placebo
- Control (Placebo Comparator): Placebo treatment will be administered for 9 days, starting on the day of ovulation triggering.
  Interventions: Drug: Resveratrol; Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — Resveratrol treatment (2 g/day) will be administered for 9 days, starting from oocyte maturation day.
  Other Names: Resverasor Plus
Drug: Placebo — Placebo treatment (2 g/day) will be administered for 9 days, starting from oocyte maturation day.

SUMMARY:
Evaluation of resveratrol treatment oh ovarian hyperstimulation syndrome in egg donors

DETAILED DESCRIPTION:
Randomized clinical trial to evaluate the role of resveratrol in preventing ovarian hyperstimulation syndrome by reducing VGEF expression and estradiol production, imporving hemoconcentration and symptomathology of this condition

ELIGIBILITY:
Inclusion Criteria:

* Number of follicles greater than 12 mm after ovarian stimulation
* Number of retrieved oocytes greater than 21

Exclusion Criteria:

* >35 years-old
* PCOS
* Endometriosis
* Systemic pathology
* Positive serologies for HBV, HBC and HIV
* Abnormal karyotype

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Serum VEGF levels | 1 day
  Serum determination of VEGF levels

SECONDARY OUTCOMES:
Hemoconcentration | 1 day
  Volume of red blood cells measured in percentage
Serum estradiol levels | 1 day
  Serum determination of estradiol levels asessed in picograms per mililiter
Ascitis | 1 day
  Volume of liquid in Douglas pouch asessed in mililiters

CONTACTS AND LOCATIONS:
Locations (1):
- Ivi Madrid, Madrid, Spain

REFERENCES:
- [Background] Ortega I, Villanueva JA, Wong DH, Cress AB, Sokalska A, Stanley SD, Duleba AJ. Resveratrol reduces steroidogenesis in rat ovarian theca-interstitial cells: the role of inhibition of Akt/PKB signaling pathway. Endocrinology. 2012 Aug;153(8):4019-29. doi: 10.1210/en.2012-1385. Epub 2012 Jun 19. PMID 22719052
- [Background] Ortega I, Wong DH, Villanueva JA, Cress AB, Sokalska A, Stanley SD, Duleba AJ. Effects of resveratrol on growth and function of rat ovarian granulosa cells. Fertil Steril. 2012 Dec;98(6):1563-73. doi: 10.1016/j.fertnstert.2012.08.004. Epub 2012 Sep 6. PMID 22959450
- [Background] Basini G, Tringali C, Baioni L, Bussolati S, Spatafora C, Grasselli F. Biological effects on granulosa cells of hydroxylated and methylated resveratrol analogues. Mol Nutr Food Res. 2010 Jul;54 Suppl 2:S236-43. doi: 10.1002/mnfr.200900320. PMID 20140899